CLINICAL TRIAL: NCT01735591
Title: An Attempt to Optimize the Results of Liver Transplantation With Administration of Probiotics.
Brief Title: Administration of Probiotics in Cirrhotic Patients Listed for Liver Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Warsaw (Other)
Collaborators: Ministry of Science and Higher Education, Poland (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 1WB/3DG1
Record Dates: First submitted 2012-11-23; First posted 2012-11-28 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2015-11

CONDITIONS: Liver Cirrhosis
Keywords: Liver cirrhosis; Liver transplantation; Probiotics; Mortality; Liver function; Infections
MeSH Terms: conditions — Liver Cirrhosis; Infections | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Probiotic (Experimental): Capsules with 3x10^9 colony forming units (Lactococcus lactis PB 411 - 50%; Lactobacillus casei PB 121 - 25%; Lactobacillus acidophilus PB 111 - 12,5%; Bifidobacterium bifidum PB 211 - 12,5%). 1 capsule a day from inclusion until liver transplantation
  Interventions: Dietary Supplement: Probiotic
- Placebo (Placebo Comparator): Placebo, 1 capsule a day from inclusion until the date of liver transplantation
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Placebo — Placebo, 1 capsule a day from inclusion until the date of liver transplantation
  Arms: Placebo
Dietary Supplement: Probiotic — Capsules with 3x10^9 colony forming units of: Lactococcus lactis PB 411 (50%), Lactobacillus casei PB 121 (25%), Lactobacillus acidophilus PB 111 (12,5%), Bifidobacterium bifidum PB 211 (12,5)
  Arms: Probiotic

SUMMARY:
The aim of this study was to evaluate the impact of the administration of probiotics on outcomes of patients qualified for liver transplantation, both in the pre-transplant period and in the early postoperative period.

DETAILED DESCRIPTION:
Gut microflora plays an important role in the pathogenesis of complications of liver cirrhosis, mainly due to microbial translocation. According to several studies, administration of probiotics in patients with cirrhosis has positive effect on minimal hepatic encephalopathy. The aim of this study was to evaluate the impact of probiotics administration on outcomes of patients qualified for liver transplantation, both in the pre-transplant period and in the early postoperative period. This study will be performed on 200 patients randomized into the probiotic and placebo groups. Daily administration of either probiotics or placebo will be continued from the date of inclusion in the study until the date of liver transplantation. A quantitative and qualitative analyses of faecal microflora will be performed in each patient before and after 10 week period (or shorter, depending on the time on the waiting list) of administration of either probiotic or placebo. Microbiological analyses of air samples from patients' home environment will be performed in each case. Both groups of patients will be compared with respect to primary and secondary outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Liver cirrhosis
* Active status on the waiting list for liver transplantation
* Confirmed etiology of liver disease

Exclusion Criteria:

* Malignancy
* Human Immunodeficiency Virus infection
* Immunosuppressive treatment prior to liver transplantation
* Cystic fibrosis
* Creatinine clearance rate < 50 mL/min

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2012-11; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
All-cause postoperative mortality | 90 days after the date of liver transplantation
Postoperative infection | 30 days from the date of liver transplantation

SECONDARY OUTCOMES:
Mortality on the waiting list | From the date of inclusion until the date of liver transplantation
Infections in the pre-transplantation period | From the date of inclusion until the date of transplantation
Primary non-function after liver transplantation | 14 days after the date of liver transplantation
Changes in model for end-stage liver disease score | From the date of inclusion until the date of transplantation
Changes in Child-Turcotte-Pugh class | From the date of inclusion until the date of transplantation
Number of hospital admissions due to infections in the pre-transplantation period | From the date of inclusion until the date of transplantation
Number of hospital admission due to complications of liver cirrhosis in the pre-transplantation period | From the date of inclusion until the date of transplantation
Serum activity of transaminases on the first 5 postoperative days | 5 days after the date of liver transplantation
Serum bilirubin concentration in the first 5 postoperative days | 5 days after the date of liver transplantation
International normalized ratio values during the first 5 postoperative days | 5 days after the date of liver transplantation
Change in model for end-stage liver disease score in the pre-transplantation period | 10 weeks
  To be assessed if the period between inclusion in the study and liver transplantation would not be shorter than 10 weeks
Change in Chil-Turcotte-Pugh class in the pre-transplantation period | 10 weeks
  To be assessed if the period between inclusion in the study and liver transplantation would not be shorter than 10 weeks

OTHER OUTCOMES:
Changes in faecal microflora | 10 weeks
  Differences in the number of colony forming units in 1 g of stool for particular bacterial and fungal species after 10 weeks of probiotic/placebo administration

CONTACTS AND LOCATIONS:
Overall Officials: Michał Grąt, M.D., Principal Investigator — Medical University of Warsaw, Department of General, Transplant and Liver Surgery; Marek Krawczyk, Professor, Study Chair — Medical University of Warsaw, Department of General, Transplant and Liver Surgery
Locations (1):
- Department of General, Transplant and Liver Surgery, Medical University of Warsaw, Warsaw, Masovian Voivodeship, Poland

REFERENCES:
- [Derived] Cooper TE, Khalid R, Chan S, Craig JC, Hawley CM, Howell M, Johnson DW, Jaure A, Teixeira-Pinto A, Wong G. Synbiotics, prebiotics and probiotics for people with chronic kidney disease. Cochrane Database Syst Rev. 2023 Oct 23;10(10):CD013631. doi: 10.1002/14651858.CD013631.pub2. PMID 37870148
- [Derived] Cooper TE, Scholes-Robertson N, Craig JC, Hawley CM, Howell M, Johnson DW, Teixeira-Pinto A, Jaure A, Wong G. Synbiotics, prebiotics and probiotics for solid organ transplant recipients. Cochrane Database Syst Rev. 2022 Sep 20;9(9):CD014804. doi: 10.1002/14651858.CD014804.pub2. PMID 36126902
- [Derived] Grat M, Grat K, Krawczyk M, Lewandowski Z, Krasnodebski M, Masior L, Patkowski W, Zieniewicz K. Post-hoc analysis of a randomized controlled trial on the impact of pre-transplant use of probiotics on outcomes after liver transplantation. Sci Rep. 2020 Nov 17;10(1):19944. doi: 10.1038/s41598-020-76994-3. PMID 33204004
- [Derived] Grat M, Wronka KM, Lewandowski Z, Grat K, Krasnodebski M, Stypulkowski J, Holowko W, Masior L, Kosinska I, Wasilewicz M, Raszeja-Wyszomirska J, Rejowski S, Bik E, Patkowski W, Krawczyk M. Effects of continuous use of probiotics before liver transplantation: A randomized, double-blind, placebo-controlled trial. Clin Nutr. 2017 Dec;36(6):1530-1539. doi: 10.1016/j.clnu.2017.04.021. Epub 2017 May 4. PMID 28506447